CLINICAL TRIAL: NCT00097968
Title: An Open-Label, Single Arm, Pilot Study of the Renal Safety of Everolimus in Addition to Neoral® in Cardiac Transplant Recipients With Established Allograft Vasculopathy
Brief Title: Safety/Efficacy of Everolimus and Neoral® in Adult Cardiac Transplant Patients With Established Allograft Vasculopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2405; RAD/Certican
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Graft Rejection
Keywords: transplant, heart, adult, everolimus; allograft rejection
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
Everolimus is an immunosuppressive drug that is being studied for preventing acute rejection that can happen after heart transplantation.

It is usually used in combination with other immunosuppressive drugs such as cyclosporine. The purpose of this study is to evaluate the change in kidney function after beginning everolimus, while determining the most effective Neoral® (cyclosporine) dose to take with everolimus, in adult cardiac transplant patients who have had their transplanted heart for at least 1 year and who have cardiac allograft vasculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult with an established cardiac allograft vasculopathy defined as any new luminal irregularity on coronary angiography.
* Patient must be on statins at study entry.
* Patient who is more than 12 months post-transplant.

Exclusion Criteria:

* Patient with a serum creatinine value >2.0 mg/dL.
* Patient with a biopsy-proven acute rejection episode (>= ISHLT 3A) within 6 months prior to study entry.
* Patient who had received any investigational drug within 4 weeks prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change in renal function at 6 assessed by comparing serum creatinine levels at 6 months to baseline values.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events at 3 and 6 months.
Patient survival at 3 and 6 months.
Treated acute rejection at 3 and 6 months.
Admission to the hospital at 3 and 6 months.
Premature study treatment discontinuation at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dorent, MD, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - University of Minnesota, Fairfield University Hospital, Minneapolis, Minnesota
  - Columbia Presbyterian Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Midstate Cardiology, Nashville, Tennessee